CLINICAL TRIAL: NCT00110175
Title: Improvement of Motor Performance in Chronic Stroke Patients by Combined Transcranial DC Stimulation and Somatosensory Stimulation
Brief Title: Motor Performance in Chronic Stroke Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050149; 05-N-0149
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-27

CONDITIONS: Stroke
Keywords: Cortical Reorganization; Motor Function; Somatosensory Stimulation; Rehabilitation; Transcranial Direct Current Stimulation (tDCS); Direct Current Stimulation; Stroke; Healthy Volunteer
MeSH Terms: conditions — Stroke

SUMMARY:
This study will determine in stroke patients whether stimulation of the injured side of the brain combined with stimulation of the weak hand can temporarily improve motor function of the paralyzed hand. It will also examine whether stimulation of the healthy side of the brain combined with stimulation of the weak hand can temporarily improve motor function in the paralyzed hand.

Healthy adult volunteers and adults who have had a stroke more than 3 months before entering the study may be eligible to participate. Candidates are screened with a physical and neurological examination. Stroke patients also have magnetic resonance imaging (MRI), a test that uses a strong magnetic field and radio waves to obtain images of the brain.

Participants perform several tasks (described below) in a practice session and then during five more sessions on separate days. They perform the tasks before and after undergoing transcranial direct current stimulation (tDCS) plus electrical stimulation (ES), and during a procedure that involves sham stimulation. For tDCS, small rubber electrodes are soaked with water and taped to the subject's head, one above the eye and the other on the back of the head. The current passes between the two electrodes. For ES, two pairs of electrodes are attached to the subject's wrist with a paste. A very short pulse of current is passed between the electrodes, creating an electrical field that stimulates the brain. For the sham stimulation, the electrodes are similarly placed, but there is no stimulation. The tasks are:

* Jebsen-Taylor test: Subjects write, lift small common objects like paper clips, and perform activities like turning pages, stacking checkers or lifting large objects. They do these tasks as fast as possible.
* Pinch force: Subjects press a wedged instrument between their thumb and index finger as hard as they can. There are several trials every 10 seconds.
* Speed tapping: Subjects press a key on a keyboard as quickly as possible for 10 seconds.
* Simple reaction time task: Subjects perform a quick wrist movement as quickly as possible in response to a "go" signal presented on a computer monitor. Muscle activity in the forearm is recorded using electrodes.
* Motor sequence learning/Learning a finger movement sequence: Subjects practice a finger movement exercise on a keyboard by pressing keys that correspond to a number displayed on a video screen.
* Visual analog scales: Subjects complete three questionnaires about their attention, fatigue, and mood.
* Sensory monitoring: Subjects are blindfolded and asked to judge the difference in various sensations, such as the feel of plastic domes with gratings, vibration, or a plastic hair applied to their fingertip.
* Scoring MRC scale: The muscle strength of the subject's hands is measured.
* Fugl-Meyer scale: The subject's ability to move his or her limbs is measured.
* Mini-mental state examination: The subject's mental ability is measured briefly.
* Handedness questionnaire: The subject's dominant hand is determined.

Participants also undergo transcranial magnetic stimulation (TMS) and electromyography (EMG) before, during and after these activities. For TMS, a wire coil is held on the scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The effect of TMS on the muscles is detected with small electrodes taped to the skin of the arms or legs. EMG measures the electrical activity of the muscles. For this test, small electrodes are taped to the skin over the muscle.

DETAILED DESCRIPTION:
There is no universally accepted strategy to promote recovery of motor function after chronic stroke, the main cause of long-term disability among adults. It is desirable to develop strategies to improve motor function in stroke patients. Recently a study in stroke patients demonstrated that transcranial direct current cortical stimulation (tDCS) in association with motor training leads to improvements of performance and motor learning. Similarly, somatosensory stimulation (peripheral nerve stimulation, PNS) of the paretic hand in stroke patients results in improvement of performance and motor learning (Celnik, unpublished data).

Objective:

The purpose of this protocol is to apply tDCS to the motor cortex of the affected hemisphere (tDCS affected) in combination with PNS of the paretic hand of patients with chronic stroke, to test the hypothesis that combined tDCS affected with PNS will lead to more prominent improvement in motor performance of functional relevant tasks in the paretic hand relative to either intervention alone.

Furthermore, recent studies have demonstrated that the unaffected hemisphere exerts abnormally high inhibitory influence over the affected hemisphere. This abnormality might adversely influence motor recovery. Therefore a further purpose of the study is to apply tDCS to the unaffected hemisphere (tDCS unaffected) to test the hypothesis that down regulation of activity in the intact hemisphere, in combination with PNS of the affected hemisphere, will elicit more prominent improvement in functional relevant tasks than either intervention alone.

Study population:

We plan to study patients with chronic strokes and healthy age, gender and hand dominance matched volunteers.

Design:

To test the hypothesis each subject will participate in 13 sessions in a double blind design. The order that patients and controls will receive the interventions will be randomized.

Outcome measures:

Primary outcome measure will be the total time to complete functional relevant tasks of the hand, Jebsen-Tailor-Test (JTT). Secondary outcomes are tapping speed with one finger; simple reaction times (SRT); pinch force; and number of correct keyboard piano sequences played in 30sec with the paretic hand. To better understand the mechanisms underlying the proposed behavioral gains, we will use transcranial magnetic stimulation (TMS) to identify corticomotor excitability changes.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include patients with thromboembolic non-hemorrhagic hemispheric lesions at least 6 months after the stroke. We will choose patients who initially had a severe motor paresis (below MRC grade 2), which subsequently recovered to the point that they have a residual motor deficit but can perform the required tasks. Assessment of the initial functional state will be taken either from patient report or medical records. As a control group, we will include age- and gender matched healthy volunteers with matched non-dominant/dominant hand (to the affected hand of the stroke patients).

EXCLUSION CRITERIA:

Patients with more than one stroke in the medial cerebral artery territory.

Patients with bilateral motor impairment.

Patients with cerebellar or brainstem lesions.

Patients or healthy volunteers unable to perform the task (wrist or elbow flexion at least MRC grade 2).

Patients or healthy volunteers with history of severe alcohol or drug abuse, psychiatric illness like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score of 23 or less).

Patients or healthy volunteers with severe uncontrolled medical problems (e.g. cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others).

Patients or healthy volunteers with increased intracranial pressure as evaluated by clinical means.

Patients with unstable cardiac arrhythmia.

Patients or healthy volunteers with h/o hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system.

Patients or healthy volunteers with more than moderate to severe microangiopathy, polyneuropathy, diabetes mellitus, or ischemic peripheral disease.

Patients or healthy volunteers with diseased or damaged skin over the face or scalp.

Patients or healthy volunteers who have professionally practiced playing a keyboard musical instrument or trained as a typist.

Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-04-28; Study Completion 2008-03-27

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Muellbacher W, Richards C, Ziemann U, Wittenberg G, Weltz D, Boroojerdi B, Cohen L, Hallett M. Improving hand function in chronic stroke. Arch Neurol. 2002 Aug;59(8):1278-82. doi: 10.1001/archneur.59.8.1278. PMID 12164724